CLINICAL TRIAL: NCT01268956
Title: Correlation of Circulating Lymphatic Progenitor Cells With Lymph Node Metastasis in Ovarian Cancer Patients
Brief Title: Circulating Lymphatic Progenitor Cell and Lymph Node Metastasis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Huiling Qiu, Department of Obstetrics & Gynecology, Southwest Hospital
Other Study IDs: 20101231001
Record Dates: First submitted 2011-01-03; First posted 2011-01-04 (Estimated); Last update posted 2011-01-04 (Estimated); Status verified 2010-12

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Lymphatic progenitor cell: Circulating lymphatic progenitor cell
- Control: healthy people

SUMMARY:
Correlation of circulating lymphatic endothelial progenitor cells with lymph node metastasis

DETAILED DESCRIPTION:
Correlation of circulating lymphatic endothelial progenitor cells with lymph node metastasis in ovarian cancer patients

ELIGIBILITY:
Inclusion Criteria:

* ovarian cancer patients diagnosed by pathologic examination

Exclusion Criteria:

* other malignant disease inflammatory disease untreated diabetic and hypertension chronic renal failure rheumatoid arthritis

Ages: 15 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: ovarian cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-06 (Estimated); Study Completion 2011-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Pianyifan pianyifan, Doctor, Principal Investigator — Southwest Hospital, China
Locations (1):
- Department of Obstetrics & Gynecology, Southwest Hospital, Chongqing, Sichuan, China